CLINICAL TRIAL: NCT00705614
Title: Crohn's Disease European Registry. A Prospective, Observational, Postmarketing Safety Surveillance Registry of Patients Treated With Remicade® or Standard Therapy
Brief Title: Postmarketing Safety Surveillance European Registry of Crohn's Disease Patients Treated With Remicade or Standard Therapy (MK-2155-035)
Acronym: ENCORE
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P03164
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Remicade Group: Particpiants with no prior exposure to Remicade, who at the time of enrollment are scheduled to receive Remicade within 30 days of the Baseline Visit. Participants who start on Remicade will constitute the Remicade Group, regardless of whether they continue with Remicade or switch to another treatment.
  Interventions: Biological: Remicade
- Standard Therapy Group: Participants who are being treated with standard therapy and are not adequately maintained and will be offered an alternative treatment that does not include Remicade. Standard therapy participants must not have previously received Remicade.
- Switched to Remicade Group: Participants who started in the Standard Therapy Group but switched over to Remicade sometime during the follow-up period. Participants who switch to Remicade are evaluated in the Standard Therapy group until the time of the switch and are evaluated in the Switched to Remicade group thereafter.
  Interventions: Biological: Remicade

INTERVENTIONS:
Biological: Remicade — The treating physician will determine the treatment regimen and dose of Remicade.
  Other Names: Infliximab; SCH 215596
  Groups: Remicade Group; Switched to Remicade Group

SUMMARY:
Prospective, observational, parallel-group, postmarketing safety surveillance registry in participants treated with Remicade or standard therapy for active or fistulizing Crohn's disease (CD). The follow-up period is up to 5 years. The participants in the standard therapy group may switch over to Remicade any time during the follow-up period

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, of either sex, and of any race.
* Must have active or fistulizing CD and must have experienced at least 1 of the following:

  * failed a tapering regimen of corticosteroids and will be initiating immunosuppressive therapy
  * required corticosteroid treatments for the previous 6 months and will be initiating immunosuppressive therapy
  * luminal or fistulizing CD, which, in the treating physician's judgment, qualifies for initiation of Remicade.
* Willing to give written informed consent and must be able to adhere to the procedural requirements of the registry.
* Must be evaluated for active and inactive (latent) tuberculosis (TB) at the Baseline Visit. TB evaluation will consist of TB history questions (eg, medical history, possible previous contact with TB, TB vaccination history). TB evaluation and TB screening (eg, skin test, chest x-ray) are required when a subject starts treatment with Remicade. In these cases, subjects must be screened for TB within 3 months prior to initiating Remicade treatment.

Exclusion Criteria:

* Female who is pregnant or nursing.
* Treated with Remicade prior to Baseline.
* Previously treated with other tumor necrosis factor (TNF)-active agents and other investigational drugs for CD prior to Baseline.
* Active or untreated latent TB or other severe infections such as sepsis, abscesses, or opportunistic infections.
* Moderate or severe heart failure (New York Heart Association [NYHA] Class III: subjects with marked limitation of activity; they are comfortable only at rest/Class IV: subjects who should be at complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest).
* Have lymphoproliferative disorders (eg, lymphoma) or malignancies.
* In a situation or have any condition that, in the opinion of the treating physician, may interfere with their optimal participation in the registry.
* Are participating in any other clinical trials (excluding registries).

In addition, subjects will be excluded from treatment with Remicade if any of the criteria listed below are met:

* Females of childbearing potential unwilling to use a medically accepted method of birth control during treatment with Remicade and to continue its use for at least 6 months after the last Remicade treatment.
* History of hypersensitivity to murine proteins or to any excipients of Remicade formulation (sucrose, polysorbate 80, monobasic sodium phosphate, and dibasic sodium phosphate).
* Other conditions that are contraindicated in the Remicade Summary of Product Characteristics (SPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects, ages 18 years and older, with a diagnosis of active or fistulizing CD with no previous exposure to Remicade will be eligible to enroll into the registry.
Sampling Method: Non-Probability Sample
Enrollment: 2662 (Actual)
Dates: Start 2003-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

REFERENCES:
- [Result] D'Haens G, Reinisch W, Colombel JF, Panes J, Ghosh S, Prantera C, Lindgren S, Hommes DW, Huang Z, Boice J, Huyck S, Cornillie F; ENCORE investigators. Five-year Safety Data From ENCORE, a European Observational Safety Registry for Adults With Crohn's Disease Treated With Infliximab [Remicade(R)] or Conventional Therapy. J Crohns Colitis. 2017 Jun 1;11(6):680-689. doi: 10.1093/ecco-jcc/jjw221. PMID 28025307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Standard Therapy group includes both those who stayed on Standard Therapy and those who switched to Remicade after starting on Standard Therapy. Two hundred ninety-eight of the 1121 subjects enrolled in the Standard Therapy Group switched to Remicade during follow-up.
Groups:
- Remicade: Participants with no prior exposure to Remicade, who at the time of enrollment, were scheduled to receive Remicade within 30 days of the enrollment visit. The treating physician will determine the treatment regimen and dose of Remicade.
- Standard Therapy Group: Participants who were treated with conventional therapies and who were adequately maintained were offered an alternative treatment that did not include Remicade. These participants must not have received treatment with Remicade prior to enrollment.
  Some participants who start in the Standard Therapy Group switched over to Remicade sometime during the follow-up period. Participants who switched to Remicade were evaluated in the Standard Therapy group until the time of the switch and were evaluated in the Switched to Remicade group thereafter.
Period: Initial Intervention
Arm/Group | Remicade | Standard Therapy Group
Started | 1541 | 1121
Completed | 1023 | 800
Not Completed | 518 | 321
Not completed — Adverse Event | 40 | 21
Not completed — Lost to Follow-up | 310 | 191
Not completed — Withdrawal by Subject | 114 | 71
Not completed — Administrative Reason | 51 | 38
Not completed — Status completion unknown | 3 | 0
Period: Switch to Remicade
Arm/Group | Remicade | Standard Therapy Group
Started | 0 | 298
Completed | 0 | 249
Not Completed | 0 | 49
Not completed — Adverse Event | 0 | 5
Not completed — Lost to Follow-up | 0 | 23
Not completed — Withdrawal by Subject | 0 | 12
Not completed — Administrative Reason | 0 | 9

BASELINE CHARACTERISTICS:
Population: 298 of the 1121 participants enrolled in the Standard Therapy Group switched to Remicade during follow-up. They are included in both the Standard Therapy and Switched to Remicade treatment groups, but baseline measures (obtained at the time of their switch to Remicade) are shown as separate rows in the Baseline Measures table.
Groups:
- Standard Therapy Group: The Standard Therapy group includes both those who stayed on Standard Therapy and those who switched to Remicade after starting on Standard Therapy. Two hundred ninety-eight of the 1121 subjects enrolled in the Standard Therapy Group switched to Remicade during follow-up.
- Total: Total of all reporting groups
Arm/Group | Remicade | Standard Therapy Group | Total
Number analyzed (Participants) | 1541 | 1121 | 2662
Age, Continuous [Mean (Standard Deviation); unit: Years]
  All Participants | 36.1 (12.90) | 37.5 (12.86) | 36.7 (12.90)
  Switched to Remicade | NA (NA) — Not available (N/A) because there are no participants in this group. | 36.7 (12.3) | 36.7 (12.3)
Sex/Gender, Customized [Number; unit: Participants]
  Female (All Participants) | 935 | 677 | 1612
  Male (All Participants) | 606 | 444 | 1050
  Female (Switched to Remicade) | NA — Not available (N/A) because there are no participants in this group. | 191 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male (Switched to Remicade) | NA — Not available (N/A) because there are no participants in this group. | 107 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Infections
Description: The number of participants experiencing serious infections was evaluated. Serious infections included, but were not limited to, tuberculosis, opportunistic infections (such as Pneumocystis carinii [PCP] pneumonia, listeriosis, atypical mycobacteria, and histoplasmosis), salmonellosis,and serious viral infections.
Time Frame: Up to 5 Years
Population: The population consisted of all enrolled participants. The Standard Therapy group was assessed only as long as they were on Standard Therapy without Remicade and the Switched group was assessed starting at the time of the switch to Remicade.
Measure: Number; unit: Participants
Groups:
- Remicade: Participants with no prior exposure to Remicade, who at the time of enrollment, were scheduled to receive Remicade within 30 days of the enrollment visit.
- Standard Therapy: Participants who were treated with conventional therapies and who were adequately maintained were offered an alternative treatment that did not include Remicade. These participants must not have received treatment with Remicade prior to enrollment.
- Switched to Remicade: Participants who started in the Standard Therapy Group but switched over to Remicade during the study.
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Participants | 132 | 47 | 18

2. Primary Outcome: Number of Participants With Infusion-Related Reactions/Hypersensitivity
Description: The number of participants with infusion-related reactions and/or hypersensitivity was evaluated. An infuson-related reaction/hypersensitivity was defined as as an acute reaction, including anaphylactic shock that occurs after the onset of the infusion or within the 1- to 2-hour observation period following the end of the infusion. Delayed hypersensitivity reactions (myalgia and/or arthralgia with fever and rash within 14 days of the infusion) were included.
Time Frame: Up to 5 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Participants | 173 | 1 | 28

3. Primary Outcome: Number of Participant Fatalities
Description: The number of participant fatalities was evaluated throughout the study.
Time Frame: Up to 5 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Participants | 30 | 14 | 4

4. Primary Outcome: Number of Participants With New or Worsening Congestive Heart Failure
Description: The number of participants with new or worsening congestive heart failure was evaluated throughout the study.
Time Frame: Up to 5 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Participants | 1 | 1 | 0

5. Primary Outcome: Number of Participants With Demyelinating Neurological Disorders
Description: The number of participants with demyelinating neurological disorders was evaluated. Demyelinating neurological disorders were defined as multiple sclerosis, optic neuritis, peripheral syndromes such as peripheral neuropathy, mononeuropathy multipex, cranial neuropathies, Guillain-Barré syndrome, chronic inflammatory demyelinating polyradiculoneuropathy, and transverse myelitis.
Time Frame: Up to 5 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Participants | 4 | 1 | 0

6. Primary Outcome: Number of Participants With Hematologic Conditions
Description: The number of participants wtih hematologic conditions was evaluated. A hematologic condition was defined as thrombocytopenia, neutropenia, pancytopenia, granulocytopenia, leukopenia, or aplastic anemia.
Time Frame: Up to 5 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Participants | 50 | 11 | 7

7. Primary Outcome: Number of Participants With Lymphoproliferative Disorders/Malignancies
Description: The number of participants wtih lymphoproliferative disorders and/or malignancies was evaluated. A lymphoproliferative disorder and /or malignancy included, but was not limited to, lymphoma, gastrointestinal cancer, skin cancer (including basocellular and squamous carcinoma, melanoma) and in situ cervical carcinoma.
Time Frame: Up to 5 Years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Participants | 49 | 21 | 8

8. Secondary Outcome: Participant Assessment of Overall Health Status By Study Visit
Description: The participant assessment of overall health status was evaluated at baseline and each study visit. The overall health status questionnaire asked participants to rate their current health status over the prior 24 hours as 1=best possible, 2=much better than average, 3=better than average, 4=average, 5=worse than average, 6=much worse than average, or 7=worst possible. Scores ranged from 1 to 7 with lower scores indicating better health status.
Time Frame: Up to 5 Years
Population: The population consisted of all enrolled participants with a Participant Assessment of Overall Health Index score at baseline and each time point. The Standard Therapy group was assessed only as long as they were on Standard Therapy without Remicade and the Switched group was assessed starting at the time of the switch to Remicade.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Score on a Scale
  Visit 1 (Baseline; n=1526, 1116, 0) | 4.3 (1.33) | 3.9 (1.38) | NA (NA) — Due to the study design, participants would not have switched to Remicade at the Baseline visit.
  Visit 2 (n=1344, 903, 95) | 3.3 (1.44) | 3.3 (1.44) | 3.9 (1.49)
  Visit 3 (n=1280, 809, 146) | 3.2 (1.41) | 3.1 (1.40) | 3.6 (1.41)
  Visit 4 (n=1217, 755, 162) | 3.2 (1.43) | 3.0 (1.38) | 3.5 (1.45)
  Visit 5 (n=1160, 704, 184) | 3.1 (1.44) | 3.1 (1.42) | 3.2 (1.52)
  Visit 6 (n=1110, 649, 202) | 3.1 (1.43) | 3.0 (1.41) | 3.4 (1.44)
  Visit 7 (n=1046, 606, 212) | 3.1 (1.47) | 3.0 (1.41) | 3.3 (1.42)
  Visit 8 (n=1044, 573, 221) | 3.1 (1.46) | 3.0 (1.44) | 3.2 (1.43)
  Visit 9 (n=999, 544, 223) | 3.1 (1.45) | 2.9 (1.41) | 3.2 (1.50)
  Visit 10 (n=963, 520, 227) | 3.0 (1.42) | 2.8 (1.44) | 3.1 (1.38)
  Visit 11 (n=956, 527, 235) | 3.0 (1.41) | 2.8 (1.43) | 3.1 (1.47)

9. Secondary Outcome: The Harvey-Bradshaw Index of Crohn's Disease Activity By Study Visit
Description: The Harvey-Bradshaw Index of Crohn's Disease Acitivity was evaluated at each study visit. The Harvey-Bradshaw Index evaluates participants' general health in the day prior in the domains of well being, abdominal pain, number of liquid stools per day, and abdominal mass and complications and was evaluated on the day of the study visit. The score is derived from a 0-4 score for general well being, 0-3 for abdmonial pain, raw score for number of liquid stools per day, 0-3 for abdominal mass, and raw score for complications. The total score is from 0 to infinity, with lower scores indicating better outcomes.
Time Frame: Up to 5 Years
Population: The population consisted of all enrolled participants with a Harvey-Bradshaw Index of Crohn's Disease score at baseline and each time point. The Standard Therapy group was assessed only as long as they were on Standard Therapy without Remicade and the Switched group was assessed starting at the time of the switch to Remicade.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Score on a Scale
  Visit 1 (Baseline; n=1505, 1106, 0) | 8.2 (5.36) | 6.2 (4.94) | NA (NA) — Due to the study design, participants would not have switched to Remicade at the Baseline visit.
  Visit 2 (n=1320, 876, 91) | 4.1 (4.13) | 3.8 (3.84) | 6.0 (5.28)
  Visit 3 (n=1250, 785, 143) | 3.7 (3.87) | 3.5 (3.64) | 4.4 (4.05)
  Visit 4 (n=1196, 742, 159) | 3.8 (4.01) | 3.2 (3.56) | 4.8 (4.47)
  Visit 5 (n=1127, 692, 181) | 3.7 (3.95) | 3.4 (3.51) | 4.9 (5.81)
  Visit 6 (n=1070, 647, 199) | 3.6 (4.00) | 3.1 (3.39) | 4.5 (4.29)
  Visit 7 (n=1023, 592, 209) | 3.6 (4.00) | 3.0 (3.36) | 4.1 (4.43)
  Visit 8 (n=1015, 562, 224) | 3.6 (3.97) | 3.2 (3.63) | 4.1 (4.69)
  Visit 9 (n=953, 546, 219) | 3.6 (4.50) | 2.9 (2.90) | 4.4 (5.23)
  Visit 10 (n=936, 526, 225) | 3.4 (4.23) | 2.7 (3.38) | 4.3 (4.66)
  Visit 11 (n=918, 525, 238) | 3.4 (3.93) | 2.7 (3.44) | 4.2 (4.29)

10. Secondary Outcome: Work/Daily Activity Status Score By Study Visit
Description: The participant work/daily activity status score was evaluated at each study visit. The work/daily activity questionnaire asked participants to rate their level of daily functioning on a scale of 1 to 10 with a lower score indicating less of an impact of Crohn's disease on work or daily life functioning.
Time Frame: Up to 5 Years
Population: The population consisted of all participants with a work/daily activity status score at baseline and each study visit. The Standard Therapy group was assessed only as long as they were on Standard Therapy without Remicade and the Switched group was assessed starting at the time of the switch to Remicade.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Score on a Scale
  Visit 1 (Baseline; n=1496, 1108, 0) | 5.9 (2.61) | 4.9 (2.83) | NA (NA) — Due to the study design, participants would not have switched to Remicade at the Baseline visit.
  Visit 2 (n=1316, 895, 94) | 4.2 (2.86) | 3.7 (2.79) | 5.5 (2.81)
  Visit 3 (n=1235, 797, 143) | 3.8 (2.76) | 3.2 (2.77) | 4.8 (2.94)
  Visit 4 (n=1192, 738, 159) | 3.6 (2.79) | 2.9 (2.60) | 4.3 (2.95)
  Visit 5 (n=1128, 694, 179) | 3.4 (2.76) | 3.0 (2.63) | 4.0 (2.89)
  Visit 6 (n=1077, 638, 201) | 3.3 (2.75) | 2.7 (2.56) | 3.9 (2.87)
  Visit 7 (n=1030, 601, 207) | 3.2 (2.70) | 2.8 (2.62) | 3.6 (2.85)
  Visit 8 (n=1025, 571, 221) | 3.3 (2.75) | 2.7 (2.59) | 3.5 (2.74)
  Visit 9 (n=982, 542, 222) | 3.3 (2.75) | 2.6 (2.46) | 3.5 (2.78)
  Visit 10 (n=934, 514, 225) | 3.1 (2.66) | 2.4 (2.53) | 3.6 (2.71)
  Visit 11 (n=925, 521, 235) | 3.2 (2.67) | 2.4 (2.44) | 3.6 (2.76)

11. Secondary Outcome: Number of Participants With a Draining Fistula By Study Visit
Description: The number of participants with a draining fistula was evaluated at each study visit.
Time Frame: Up to 5 Years
Population: The population consisted of all enrolled participants with fistula status data. The Standard Therapy group was assessed only as long as they were on Standard Therapy without Remicade and the Switched group was assessed starting at the time of the switch to Remicade.
Measure: Number; unit: Participants
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Participants
  Visit 1 (Baseline; n=1541, 1120, 0) | 349 | 96 | NA — Due to the study design, participants would not have switched to Remicade at the Baseline visit.
  Visit 2 (n=1420, 920, 100) | 211 | 51 | 16
  Visit 3 (n=1334, 827, 152) | 170 | 41 | 19
  Visit 4 (n=1285, 779, 168) | 146 | 31 | 12
  Visit 5 (n=1221, 714, 188) | 125 | 29 | 15
  Visit 6 (n=1169, 666, 208) | 114 | 26 | 15
  Visit 7 (n=1110, 615, 219) | 97 | 31 | 15
  Visit 8 (n=1097, 588, 233) | 105 | 23 | 16
  Visit 9 (n=1046, 562, 229) | 98 | 32 | 15
  Visit 10 (n=1030, 535, 235) | 85 | 15 | 20
  Visit 11 (n=1006, 541, 248) | 87 | 16 | 20

12. Secondary Outcome: Number of Participant Hospital Stays for Crohn's Disease in the Prior 6 Months
Description: The number of participant hospital stays for Crohn's Disease in the prior 6 months was evaluated at each study visit.
Time Frame: Up to 5 Years
Population: The population consisted of all enrolled participants with hospital stay data. The Standard Therapy group was assessed only as long as they were on Standard Therapy without Remicade and the Switched group was assessed starting at the time of the switch to Remicade.
Measure: Mean (Standard Deviation); unit: Hospital Stays
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Hospital Stays
  Visit 1 (Baseline; n=1539, 1121, 0) | 0.7 (1.25) | 0.5 (0.81) | NA (NA) — Due to the study design, participants would not have switched to Remicade at the Baseline visit.
  Visit 2 (n=1418, 920, 100) | 0.3 (0.87) | 0.2 (0.50) | 0.5 (0.76)
  Visit 3 (n=1334, 827, 152) | 0.3 (0.92) | 0.1 (0.38) | 0.4 (0.86)
  Visit 4 (n=1285, 779, 168) | 0.2 (0.56) | 0.2 (3.08) | 0.2 (0.67)
  Visit 5 (n=1221, 714, 188) | 0.1 (0.54) | 0.1 (0.28) | 0.3 (0.72)
  Visit 6 (n=1170, 665, 208) | 0.1 (0.66) | 0.1 (0.33) | 0.1 (0.49)
  Visit 7 (n=1111, 615, 219) | 0.1 (0.40) | 0.1 (0.43) | 0.2 (0.55)
  Visit 8 (n=1099, 589, 233) | 0.1 (0.76) | 0.1 (0.42) | 0.1 (0.49)
  Visit 9 (n=1046, 562, 229) | 0.1 (0.68) | 0.1 (0.50) | 0.1 (0.31)
  Visit 10 (n=1031, 535, 235) | 0.1 (0.46) | 0.1 (0.42) | 0.1 (0.44)
  Visit 11 (n=1006, 541, 248) | 0.1 (0.35) | 0.1 (2.59) | 0.1 (0.42)

13. Secondary Outcome: Duration of Participant Hospital Stays for Crohn's Disease in the Prior 6 Months
Description: The duration of hospital stays for Crohn's Disease in the prior 6 months was evaluated at each study visit.
Time Frame: Up to 5 Years
Population: The population consisted of all enrolled participants with hospital stay duration data. The Standard Therapy group was assessed only as long as they were on Standard Therapy without Remicade and the Switched group was assessed starting at the time of the switch to Remicade.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Days
  Visit 1 (Baseline; n=657,418 ,0) | 12.2 (13.73) | 10.8 (10.93) | NA (NA) — Due to the study design, participants would not have switched to Remicade at the Baseline visit.
  Visit 2 (n=304,126, 33) | 14.4 (17.81) | 12.0 (14.26) | 13.0 (12.23)
  Visit 3 (n=216, 58, 35) | 14.2 (16.83) | 9.4 (7.49) | 13.5 (13.65)
  Visit 4 (n=151, 60, 24) | 12.6 (15.23) | 8.5 (11.87) | 9.1 (10.82)
  Visit 5 (n=105, 35, 34) | 11.7 (13.02) | 9.8 (9.49) | 7.1 (6.21)
  Visit 6 (n=107, 49, 19) | 10.8 (17.33) | 13.7 (27.34) | 18.3 (17.81)
  Visit 7 (n=109, 45, 25) | 10.6 (14.41) | 10.2 (10.63) | 10.0 (11.33)
  Visit 8 (n=98, 29, 23) | 9.5 (9.04) | 16.3 (15.52) | 14.7 (17.29)
  Visit 9 (n=80, 38, 17) | 12.4 (14.44) | 6.9 (5.77) | 10.7 (17.20)
  Visit 10 (n=85, 29, 27) | 10.1 (12.02) | 8.0 (5.41) | 9.0 (6.40)
  Visit 11 (n=63, 19, 18) | 11.4 (13.24) | 8.7 (10.64) | 18.1 (31.57)

14. Secondary Outcome: Number of Participant Surgical Procedures for Crohn's Disease in the Prior 6 Months
Description: The number of participants undergoing surgical procedures for Crohn's Disease in the prior 6 months was evaluated at each study visit.
Time Frame: Up to 5 Years
Population: The population consisted of all enrolled participants with surgical procedure data. The Standard Therapy group was assessed only as long as they were on Standard Therapy without Remicade and the Switched group was assessed starting at the time of the switch to Remicade.
Measure: Number; unit: Surgical Procedures
Arm/Group | Remicade | Standard Therapy | Switched to Remicade
Number analyzed (Participants) | 1541 | 1121 | 298
Surgical Procedures
  Visit 1 (Basline; n=660, 419, 0) | 171 | 81 | NA — Due to the study design, participants would not have switched to Remicade at the Baseline visit.
  Visit 2 (n=304, 126, 33) | 135 | 51 | 7
  Visit 3 (n=217, 57, 36) | 121 | 23 | 12
  Visit 4 (n=153, 60, 24) | 68 | 16 | 8
  Visit 5 (n=106, 36, 34) | 50 | 14 | 14
  Visit 6 (n=108, 49, 19) | 49 | 21 | 11
  Visit 7 (n=109, 45, 25) | 48 | 20 | 6
  Visit 8 (n=98, 29, 23) | 43 | 12 | 7
  Visit 9 (n=82, 38, 17) | 38 | 13 | 8
  Visit 10 (n=85, 29, 27) | 38 | 13 | 8
  Visit 11 (n=63, 19, 18) | 34 | 6 | 8

ADVERSE EVENTS:
Time Frame: Up to 5 Years
Arm/Group | Standard Therapy | Remicade | Switched to Remicade
Serious Adverse Events (participants affected / at risk) | 391/1121 | 792/1541 | 136/298
Other Adverse Events (participants affected / at risk) | 173/1121 | 441/1541 | 51/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=1121) | Remicade (N=1541) | Switched to Remicade (N=298)
ANAEMIA (Blood and lymphatic system disorders) | 5 (6) | 9 (11) | 1 (1)
ANAEMIA HAEMOLYTIC AUTOIMMUNE (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA VITAMIN B12 DEFICIENCY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THYMUS DISORDER (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (4) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
CARDIAC VALVE DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PLEUROPERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
TACHYARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CONGENITAL ANOMALY IN OFFSPRING (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
ENCEPHALOCELE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMANGIOMA CONGENITAL (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
HIP DYSPLASIA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
PRETERNATURAL ANUS (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
ADRENOCORTICAL INSUFFICIENCY ACUTE (Endocrine disorders) | 0 (0) | 1 (2) | 0 (0)
GOITRE (Endocrine disorders) | 3 (3) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
COLOUR BLINDNESS ACQUIRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
UVEITIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 7 (7) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 29 (30) | 42 (49) | 9 (10)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (4) | 5 (5) | 1 (1)
ACUTE ABDOMEN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ANAL FISSURE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
ANAL FISTULA (Gastrointestinal disorders) | 11 (18) | 47 (57) | 4 (5)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ANAL SKIN TAGS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ANAL SPHINCTER ATONY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ANAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
ANOGENITAL DYSPLASIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ANOVULVAR FISTULA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
BILE ACID MALABSORPTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 6 (6) | 8 (8) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0)
COLONIC FISTULA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
COLONIC STENOSIS (Gastrointestinal disorders) | 2 (2) | 8 (9) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 131 (164) | 298 (460) | 47 (67)
DIARRHOEA (Gastrointestinal disorders) | 6 (6) | 11 (12) | 4 (4)
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DUODENAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ENTEROCOLONIC FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 3 (6) | 7 (9) | 1 (1)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
FAECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
FAECALOMA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
FOOD POISONING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
GASTRODUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
GASTROINTESTINAL DYSPLASIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL FISTULA (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 3 (7) | 1 (1)
GASTROINTESTINAL HYPOMOTILITY (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL STENOSIS (Gastrointestinal disorders) | 7 (8) | 9 (15) | 3 (3)
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HERNIAL EVENTRATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ILEAL FISTULA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
ILEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ILEAL STENOSIS (Gastrointestinal disorders) | 20 (21) | 41 (45) | 9 (10)
ILEITIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
ILEUS (Gastrointestinal disorders) | 12 (13) | 17 (19) | 4 (5)
INFLAMMATORY BOWEL DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
INTESTINAL ANGINA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL FISTULA (Gastrointestinal disorders) | 2 (2) | 7 (7) | 1 (1)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL INFARCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 9 (10) | 36 (44) | 4 (4)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
INTESTINAL POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL STENOSIS (Gastrointestinal disorders) | 8 (8) | 15 (16) | 3 (3)
INTUSSUSCEPTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
JEJUNAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3)
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 2 (2) | 9 (9) | 1 (1)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
MALABSORPTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MECHANICAL ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
MESENTERIC OCCLUSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MESENTERIC VASCULAR INSUFFICIENCY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 7 (7) | 1 (1)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 5 (5) | 6 (8) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (4)
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
POUCHITIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 5 (7) | 0 (0)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PROCTOCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1)
RECTAL PROLAPSE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
RECTAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 8 (9) | 16 (17) | 1 (1)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
SMALL INTESTINAL STENOSIS (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
SUBILEUS (Gastrointestinal disorders) | 11 (13) | 17 (21) | 6 (7)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 4 (4) | 10 (10) | 1 (1)
ADHESION (General disorders) | 1 (1) | 1 (1) | 0 (0)
ADVERSE DRUG REACTION (General disorders) | 1 (1) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
CONDITION AGGRAVATED (General disorders) | 1 (1) | 0 (0) | 0 (0)
CYST (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEATH NEONATAL (General disorders) | 0 (0) | 1 (1) | 0 (0)
DRUG INEFFECTIVE (General disorders) | 0 (0) | 1 (1) | 0 (0)
DRUG INTOLERANCE (General disorders) | 1 (1) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 2 (2) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 4 (4) | 0 (0)
HERNIA (General disorders) | 0 (0) | 2 (2) | 1 (1)
IMPAIRED HEALING (General disorders) | 2 (2) | 3 (3) | 0 (0)
INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
LOCALISED OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0) | 2 (3)
MEDICAL DEVICE COMPLICATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 0 (0) | 1 (1) | 0 (0)
NECROSIS (General disorders) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 4 (4) | 2 (2) | 2 (2)
OEDEMA (General disorders) | 1 (1) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 3 (3) | 0 (0)
PYREXIA (General disorders) | 9 (10) | 16 (19) | 4 (4)
SEROSITIS (General disorders) | 1 (1) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (2) | 1 (1) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 3 (3) | 1 (1)
CHOLANGITIS SCLEROSING (Hepatobiliary disorders) | 1 (2) | 1 (2) | 1 (2)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 2 (3) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTOCHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 5 (5) | 8 (8) | 2 (2)
CHOLESTASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLESTASIS OF PREGNANCY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0)
HEPATORENAL FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
PORTAL HYPERTENSION (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 (1) | 2 (2) | 0 (0)
ANAPHYLACTOID REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 4 (4) | 11 (11) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 7 (7) | 0 (0)
INTESTINE TRANSPLANT REJECTION (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
SERUM SICKNESS (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
TYPE IV HYPERSENSITIVITY REACTION (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 7 (8) | 20 (23) | 2 (3)
ABDOMINAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
ABSCESS (Infections and infestations) | 10 (11) | 10 (10) | 1 (1)
ABSCESS INTESTINAL (Infections and infestations) | 1 (1) | 4 (5) | 3 (3)
ABSCESS SWEAT GLAND (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ACINETOBACTER BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ACUTE TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
AMOEBIC DYSENTERY (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 17 (21) | 61 (83) | 8 (12)
APPENDICITIS (Infections and infestations) | 3 (3) | 7 (7) | 1 (1)
ARTHRITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BARTHOLIN'S ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
CAMPYLOBACTER INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
CHLAMYDIAL INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
CHRONIC SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CHRONIC TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 5 (5) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
CYTOMEGALOVIRUS HEPATITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 5 (5) | 4 (5) | 0 (0)
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENDOCARDITIS STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 9 (9) | 16 (16) | 2 (2)
GASTROENTERITIS PSEUDOMONAS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GENITAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GENITOURINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GIARDIASIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
GROIN ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HAEMATOMA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS E (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HERPES VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 5 (5) | 1 (1)
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HORDEOLUM (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HUMAN HERPESVIRUS 6 INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTIVE THROMBOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LARYNGITIS (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
LISTERIOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
LIVER ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LOBAR PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MENINGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MENINGITIS LISTERIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MENINGITIS STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MENINGITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MENINGOENCEPHALITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MYCOBACTERIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MYCOPLASMA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OVARIAN ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PAPILLOMA VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PELVIC ABSCESS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PERINEAL ABSCESS (Infections and infestations) | 1 (1) | 4 (5) | 0 (0)
PERIRECTAL ABSCESS (Infections and infestations) | 1 (1) | 6 (6) | 0 (0)
PERITONEAL ABSCESS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (1) | 7 (8) | 1 (1)
PERITONSILLAR ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PILONIDAL CYST (Infections and infestations) | 2 (2) | 3 (4) | 0 (0)
PNEUMONIA (Infections and infestations) | 5 (5) | 14 (15) | 2 (2)
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
POSTOPERATIVE ABSCESS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PSOAS ABSCESS (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PURULENT DISCHARGE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 4 (4) | 2 (2)
RECTAL ABSCESS (Infections and infestations) | 1 (1) | 7 (8) | 0 (0)
RECTOVAGINAL SEPTUM ABSCESS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
RETROPERITONEAL ABSCESS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
SALMONELLOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SALPINGITIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
SEPSIS (Infections and infestations) | 2 (2) | 7 (7) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
STITCH ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 2 (2) | 8 (8) | 1 (1)
TONSILLITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TOXOPLASMOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
TUBERCULOSIS GASTROINTESTINAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 5 (5) | 0 (0)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VAGINAL ABSCESS (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VIRAL DIARRHOEA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VIRAL PERICARDITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
VULVAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
ANASTOMOTIC COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ANASTOMOTIC FISTULA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
EXPOSURE DURING PREGNANCY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 5 (5)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 7 (8) | 1 (2)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HEPATIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 2 (3) | 4 (4) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
POISONING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 0 (0)
POST PROCEDURAL DIARRHOEA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
POSTOPERATIVE HERNIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TENDON INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TOOTH INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
BIOPSY LIVER (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD SODIUM DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
CYTOMEGALOVIRUS TEST (Investigations) | 0 (0) | 1 (1) | 0 (0)
FALSE POSITIVE INVESTIGATION RESULT (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (2) | 0 (0)
INVESTIGATION (Investigations) | 1 (1) | 2 (2) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
NOROVIRUS TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | 0 (0)
VOLUME BLOOD DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 2 (2) | 2 (3) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 11 (27) | 3 (3)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
FLUID RETENTION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
FOOD INTOLERANCE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 1 (2)
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OVERWEIGHT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
VITAMIN K DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (11) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 0 (0)
ARTHRITIS ENTEROPATHIC (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
ARTHRITIS REACTIVE (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (7) | 0 (0)
FISTULA (Musculoskeletal and connective tissue disorders) | 6 (6) | 17 (17) | 2 (3)
FISTULA DISCHARGE (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
FRACTURE DELAYED UNION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1)
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
METATARSALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MONARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
SLE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
TRISMUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 3 (3) | 0 (0)
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0)
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BENIGN SOFT TISSUE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BENIGN UTERINE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
MALIGNANT NEOPLASM OF UNKNOWN PRIMARY SITE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT PERITONEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
METASTATIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINE ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
URETERIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 1 (1)
VULVAL CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL ARTERY THROMBOSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL ATROPHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
GRAND MAL CONVULSION (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 3 (4) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
NERVE ROOT COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OPTIC NEURITIS (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PYRAMIDAL TRACT SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
TENSION HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) | 1 (1)
BREECH PRESENTATION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
DELIVERY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) | 0 (0)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
FOETAL DISORDER (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
FOETAL GROWTH RESTRICTION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
GESTATIONAL DIABETES (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
NORMAL LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
PLACENTAL DISORDER (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
POSTPARTUM HAEMORRHAGE (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
PRE-ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) | 0 (0)
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 3 (4) | 20 (20) | 1 (1)
PREMATURE BABY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 1 (1)
PREMATURE DELIVERY (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 1 (1)
TWIN PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
UMBILICAL GRANULOMA (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
UTERINE CONTRACTIONS ABNORMAL (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
AGGRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 4 (4) | 6 (9) | 1 (1)
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DYSTHYMIC DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ENCOPRESIS (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
PANIC ATTACK (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
POST-TRAUMATIC STRESS DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SOMATISATION DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
CALCULUS URETERIC (Renal and urinary disorders) | 1 (2) | 2 (2) | 1 (1)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0)
IGA NEPHROPATHY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 5 (8) | 10 (11) | 1 (1)
PNEUMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
POSTRENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 1 (2) | 4 (5) | 1 (2)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 4 (4) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
RENAL MASS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URETERIC STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URETHRAL FISTULA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
BARTHOLIN'S CYST (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
BARTHOLINITIS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
BREAST MASS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 0 (0)
CYSTOCELE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
EPIDIDYMITIS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 3 (3) | 8 (9) | 0 (0)
INFERTILITY (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 3 (3) | 4 (4) | 0 (0)
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
OVARIAN DISORDER (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
PERINEAL FISTULA (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 0 (0)
UTERINE MALPOSITION (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
VAGINAL FISTULA (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7) | 1 (1)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE FEBRILE NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS BULLOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DYSHIDROTIC ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
HENOCH-SCHONLEIN PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
FAMILIAL RISK FACTOR (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
PREGNANCY OF PARTNER (Social circumstances) | 0 (0) | 2 (2) | 0 (0)
CAESAREAN SECTION (Surgical and medical procedures) | 1 (1) | 5 (5) | 2 (3)
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
COLECTOMY (Surgical and medical procedures) | 0 (0) | 3 (3) | 1 (1)
COLOSTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
COLOSTOMY CLOSURE (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
ENTEROSTOMY (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
FISTULA REPAIR (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
HAEMATOPOIETIC STEM CELL MOBILISATION (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
HOSPITALISATION (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
HYSTERECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
ILEECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
ILEOSTOMY (Surgical and medical procedures) | 0 (0) | 4 (4) | 0 (0)
ILEOSTOMY CLOSURE (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL ANASTOMOSIS (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL RESECTION (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
LIVER TRANSPLANT (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
MACROPHAGE ACTIVATION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
MITRAL VALVE REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
POLYPECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL RESECTION (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
SURGERY (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
THYROIDECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
AORTIC DISSECTION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC OCCLUSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ARTERIAL THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 4 (5) | 1 (1)
HAEMATOMA (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
HYPERTENSION (Vascular disorders) | 4 (4) | 2 (2) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 2 (3) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1) | 1 (2) | 0 (0)
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=1121) | Remicade (N=1541) | Switched to Remicade (N=298)
ABDOMINAL PAIN (Gastrointestinal disorders) | 41 (45) | 100 (124) | 15 (18)
CROHN'S DISEASE (Gastrointestinal disorders) | 64 (84) | 153 (195) | 19 (23)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 124 (153) | 281 (376) | 37 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall have editorial rights with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.